CLINICAL TRIAL: NCT00576823
Title: 12-week, Multicenter, Open-label, Non-comparative Study to Investigate Pharmacodynamic and Safety of Alfuzosin 0.2 mg/kg/Day in the Treatment of Children and Adolescents 2 - 16 Years of Age With Hydronephrosis Associated With Elevated Detrusor Leak Point Pressure of Neuropathic Etiology Followed by a 40-week Open-label Extension
Brief Title: Alfuzosin Treatment in Children and Adolescents With Hydronephrosis of Neuropathic Etiology
Acronym: Alfahydro
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC6269; SL770499; 2004-002397-38 (EudraCT Number)
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Results first posted 2011-02-08 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Hydronephrosis; Neurogenic Bladder
Keywords: child; bladder; neuropathic; alpha blockers
MeSH Terms: conditions — Hydronephrosis; Urinary Bladder, Neurogenic | interventions — alfuzosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alfuzosin solution - 2-7 years (Experimental): Alfuzosin solution, daily dose divided in 3 doses given at breakfast, lunch and dinner to children 2-7 years of age.
  Interventions: Drug: Alfuzosin
- Alfuzosin solution - 8-16 years (Experimental): Alfuzosin solution, daily dose divided in 3 doses given at breakfast, lunch and dinner to children and adolescents 8-16 years of age who were not able to swallow tablets or preferred to take the solution or had a body weight < 30 kg.
  Interventions: Drug: Alfuzosin
- Alfuzosin tablet - 8-16 years (Experimental): Alfuzosin tablet, daily dose divided in 2 doses given at breakfast and dinner to children and adolescents 8-16 years of age who were able to swallow tablets and had a body weight ≥ 30 kg.
  Interventions: Drug: Alfuzosin

INTERVENTIONS:
Drug: Alfuzosin — Dose: 0.2 mg/kg/day
  Route: oral
  Other Names: SL770499

SUMMARY:
Primary objective was to determine efficacy of Alfuzosin in the treatment of children and adolescents 2-16 years of age with newly diagnosed or progressive hydronephrosis due to elevated detrusor Leak Point Pressure [LPP] of neuropathic etiology.

Secondary objectives were:

* To investigate the safety and tolerability of alfuzosin 0.2 mg/kg/day in children and adolescents,
* To investigate the number of Urinary Tract Infection (UTI) episodes,
* To investigate the pharmacokinetics of Alfuzosin (population kinetics).

DETAILED DESCRIPTION:
The study consisted of 2 phases:

* a 12-week efficacy phase then,
* a 40-week safety extension phase.

All eligible subjects received alfuzosin 0.2 mg/kg/day. The formulation and the frequency was assigned by Interactive Voice Response System (IVRS) according to age group and ability to swallow tablets.

Patients who completed the 12-week open-label treatment period were offered to continue in the 40-week open-label safety extension study. The treatment was the same as in the 12-week efficacy phase.

All patients had a one-week follow-up period after the last dose intake.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents of either gender 2 - 16 years of age with a detrusor Leak Point Pressure (LPP) of 40 cm water or greater and with newly diagnosed or progressive hydronephrosis either Society of Fetal Urology (SFU) grade 1, 2 or 3 due to neuropathic bladder dysfunction.

Exclusion Criteria:

* Hydronephrosis of non-neuropathic etiology.
* Urological surgery in the last 4 months prior to the study.
* Urethral dilatation in the last 3 months prior to the baseline urodynamic assessment.
* α-blocker therapy in the last 4 weeks prior to the baseline urodynamic assessment.
* Detrusor injections of botulinum toxin in the last 6 months.
* Urological diseases/conditions other than functional bladder obstruction of neuropathic etiology, that can lead to upper urinary tract dilatation (e.g., bladder anomalies, ureterocele).
* History of intolerance to α-blocker therapy.
* Orthostatic hypotension.
* History of risk factors for Torsade de pointes (e.g., family history of Long QT Syndrome).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2007-12; Primary Completion 2009-01 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (12):
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Belgrade, Serbia
- Sanofi-Aventis Aministrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 19 sites in 12 countries. A total of 42 patients were screened between December 2007 and September 2008.
Pre-assignment Details: 18 of the 42 screened patients were not included in the study. The reasons were the following:
  * Inclusion/Exclusion criteria not respected (16 patients),
  * Subject's request (1 patient),
  * Other (2 patients).
  Patients could have several reasons for not being included.
Groups:
- Alfuzosin Solution - 8-16 Years: Alfuzosin solution, daily dose divided in 3 doses given at breakfast, lunch and dinner to children and adolescents 8-16 years of age who were not able to swallow the tablets or preferred to take the solution or had a body weight < 30 kg.
- Alfuzosin Tablet - 8-16 Years: Alfuzosin tablet, daily dose divided in 2 doses given at breakfast and dinner to children and adolescents 8-16 years of age who were able to swallow the tablets and had a body weight ≥ 30 kg.
Period: 12-week Efficacy Phase
Arm/Group | Alfuzosin Solution - 2-7 Years | Alfuzosin Solution - 8-16 Years | Alfuzosin Tablet - 8-16 Years
Started | 12 | 6 | 7
Completed | 11 | 6 | 7
Not Completed | 1 | 0 | 0
Not completed — Parent's schedule issue | 1 | 0 | 0
Period: 40-week Safety Extension Phase
Arm/Group | Alfuzosin Solution - 2-7 Years | Alfuzosin Solution - 8-16 Years | Alfuzosin Tablet - 8-16 Years
Started | 11 | 6 | 6 (One patient refused to continue in the extension phase.)
Completed | 10 | 6 | 6
Not Completed | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alfuzosin Solution - 2-7 Years | Alfuzosin Solution - 8-16 Years | Alfuzosin Tablet - 8-16 Years | Total
Number analyzed (Participants) | 12 | 6 | 7 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.3 (1.5) | 10.0 (1.7) | 11.2 (2.3) | 7.9 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 5 | 16
  Male | 5 | 2 | 2 | 9
Region of Enrollment [Number; unit: participants]
  Taiwan | 0 | 1 | 1 | 2
  Slovakia | 1 | 0 | 1 | 2
  Poland | 4 | 2 | 2 | 8
  Malaysia | 0 | 0 | 1 | 1
  Singapore | 1 | 0 | 0 | 1
  Turkey | 1 | 0 | 0 | 1
  Russian Federation | 3 | 2 | 2 | 7
  India | 2 | 1 | 0 | 3
Type of hydronephrosis [Number; unit: participants]
  Bilateral hydronephrosis (both kidneys affected) | 11 | 4 | 5 | 20
  Unilateral hydronephrosis (one kidney affected) | 1 | 2 | 2 | 5
Grade of hydronephrosis [Median (Full Range); unit: grade] — Hydronephrosis was investigated by ultrasound of the kidneys, and graded using the Society of Fetal Urology (SFU) classification [5-point ordinal scale grading hydronephrosis from 0 (No hydronephrosis) to 4 (worst condition)].
  grade
    Left kidney | 2 [1 to 3] | 1.5 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
    Right kidney | 1 [0 to 3] | 2 [0 to 3] | 1 [0 to 3] | 1 [0 to 3]
Duration of diagnosis for hydronephrosis [Mean (Standard Deviation); unit: years] | 1.83 (2.30) | 5.45 (4.20) | 3.35 (3.05) | 3.12 (3.26)
Urinary Tract Infection (UTI) history within the last 3 months [Number; unit: participants]
  No UTI episode | 9 | 4 | 6 | 19
  One UTI episode | 2 | 2 | 1 | 5
  Two UTI episodes | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Decrease From Baseline ≥ 1 in the Society of Fetal Urology (SFU) Grade of Hydronephrosis
Description: Hydronephrosis was investigated by ultrasound and graded using SFU classification at each time point.
  'Complete response' was assessed when bilateral hydronephrosis at baseline and grade decrease from baseline ≥ 1 for both kidneys, or, unilateral hydronephrosis at baseline and grade decrease from baseline ≥ 1 for the affected kidney without worsening of the other kidney.
  'Partial response' was assessed when bilateral hydronephrosis at baseline and grade decrease from baseline ≥ 1 for one kidney without worsening of the other kidney.
Time Frame: baseline and 12 weeks (efficacy study phase)
Population: The analysis was on the intent-to-treat (ITT) population (i.e. all included patients who received at least one dose of Alfuzosin) excluding the patients who didn't have baseline SFU grade. Patients without post-baseline SFU grade before Week 12 were included as non-responders.
Measure: Number; unit: participants
Arm/Group | Alfuzosin Solution - 2-7 Years | Alfuzosin Solution - 8-16 Years | Alfuzosin Tablet - 8-16 Years
Number analyzed (Participants) | 12 | 6 | 7
participants
  Complete response | 2 | 5 | 3
  - Bilateral hydronephrosis | 1 | 3 | 1
  - Unilateral hydronephrosis | 1 | 2 | 2
  Partial response | 3 | 0 | 3

2. Secondary Outcome: Number of Participants With Symptomatic Urinary Tract Infection (UTI) Episodes
Description: When a patient presented with symptoms such as pain, fever or hematuria (discretion of the Investigator), an urinalysis was performed including a dipstick and a quantitative urine culture.
  A symptomatic UTI was defined as the presence of symptoms and a positive culture with > 100 000 Colony Forming Units (CFUs) with a single organism.
Time Frame: 12 weeks (efficacy study phase)
Population: The analysis was performed on the ITT population (i.e. all included patients who received at least one dose of Alfuzosin).
Measure: Number; unit: participants
Arm/Group | Alfuzosin Solution - 2-7 Years | Alfuzosin Solution - 8-16 Years | Alfuzosin Tablet - 8-16 Years
Number analyzed (Participants) | 12 | 6 | 7
participants
  No symptomatic UTI | 11 | 5 | 7
  One symptomatic UTI | 0 | 1 | 0
  Two symptomatic UTI | 1 | 0 | 0

3. Secondary Outcome: Number of Participants With Symptomatic Urinary Tract Infection (UTI) Episodes
Time Frame: 52 weeks (efficacy and extension study phases)
Population: The analysis was performed on the exposed population (i.e. all patients who received at least one dose of Alfuzosin regardless of the amount of treatment received).
Measure: Number; unit: participants
Arm/Group | Alfuzosin Solution - 2-7 Years | Alfuzosin Solution - 8-16 Years | Alfuzosin Tablet - 8-16 Years
Number analyzed (Participants) | 12 | 6 | 7
participants
  No symptomatic UTI | 8 | 5 | 5
  One symptomatic UTI | 2 | 0 | 2
  Two symptomatic UTI | 2 | 0 | 0
  Three symptomatic UTI | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) regardless of seriousness or relationship to drug, spanning from signature of the informed consent form up to the last visit were collected.
Description: The analysis was performed on the exposed population (i.e. all included patients exposed to Alfuzosin regardless of the amount of treatment administered) and included all AE that developed/worsened during the 'on treatment period' (i.e. from first dose up to 2 days after the last dose of Alfuzosin).
Groups:
- Afluzosin Solution - 2-7 Years: Alfuzosin solution, daily dose divided in 3 doses given at breakfast, lunch and dinner to children 2-7 years of age.
- Afluzosin Solution - 8-16 Years: Alfuzosin solution, daily dose divided in 3 doses given at breakfast, lunch and dinner to children and adolescents 8-16 years of age who were not able to swallow the tablets or preferred to take the solution or had a body weight < 30 kg.
- Afluzosin Tablets - 8-16 Years: Alfuzosin tablet, daily dose divided in 2 doses given at breakfast and dinner to children and adolescents 8-16 years of age who were able to swallow the tablets and had a body weight ≥ 30 kg.
Arm/Group | Afluzosin Solution - 2-7 Years | Afluzosin Solution - 8-16 Years | Afluzosin Tablets - 8-16 Years
Serious Adverse Events (participants affected / at risk) | 2/12 | 2/6 | 0/7
Other Adverse Events (participants affected / at risk) | 9/12 | 5/6 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afluzosin Solution - 2-7 Years (N=12) | Afluzosin Solution - 8-16 Years (N=6) | Afluzosin Tablets - 8-16 Years (N=7)
PYELONEPHRITIS (Infections and infestations) | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
CONVULSION (Nervous system disorders) | 0 | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 0
CALCULUS URINARY (Renal and urinary disorders) | 1 | 0 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
URETERIC INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afluzosin Solution - 2-7 Years (N=12) | Afluzosin Solution - 8-16 Years (N=6) | Afluzosin Tablets - 8-16 Years (N=7)
CYSTITIS (Infections and infestations) | 3 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 3 | 1 | 0
PHARYNGITIS (Infections and infestations) | 1 | 1 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1
CONJUNCTIVITIS INFECTIVE (Infections and infestations) | 0 | 0 | 1
EAR INFECTION (Infections and infestations) | 1 | 0 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 0 | 0
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 0
TONSILLITIS (Infections and infestations) | 0 | 0 | 1
VIRAL INFECTION (Infections and infestations) | 1 | 0 | 0
VIRAL PHARYNGITIS (Infections and infestations) | 0 | 1 | 0
VIRAL RHINITIS (Infections and infestations) | 1 | 0 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 1
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 1 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
LEUKOCYTURIA (Renal and urinary disorders) | 1 | 0 | 0
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 1 | 0 | 0
PYREXIA (General disorders) | 2 | 2 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1 | 0
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
IATROGENIC INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
URETHRAL INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This was an exploratory, open-label, non-comparative trial. Analyses were purely descriptive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months after trial completion, the investigators can publish the results. Prior to the publication, the sponsor can review and request changes to the manuscript, provided they do not jeopardize the accuracy and/or the scientific value of the publication. The approval is given in writing by the sponsor, not to exceed 90 days.

To protect by a property right any information the sponsor can postpone the publication, for a period not to exceed 18 months.